CLINICAL TRIAL: NCT02031146
Title: Lumbar Puncture and Syphilis Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Christina Marra, Professor, Neurology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001718; R01NS082120 (NIH)
Record Dates: First submitted 2014-01-06; First posted 2014-01-09 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LP (Other): Participants undergo lumbar puncture for CSF evaluation
  Interventions: Procedure: Lumbar puncture
- No LP (No Intervention): Participants do not undergo lumbar puncture and CSF is not examined.

INTERVENTIONS:
Procedure: Lumbar puncture
  Arms: LP

SUMMARY:
Treponema pallidum, the bacterium that causes syphilis, invades the central nervous system in about 40% of patients with syphilis. This happens early after infection. Patients with neuroinvasion are at risk of developing serious neurological complications, including vision or hearing loss, stroke and dementia. Because neuroinvasion can happen without symptoms, the only way to identify it is by performing a lumbar puncture (LP) to examine cerebrospinal fluid (CSF).The overall hypothesis to be tested in this study is that a strategy of immediate LP, followed by therapy based on CSF evaluation, results in better serological and functional outcomes in patients with syphilis who are at high risk for neuroinvasion.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18 years or older
2. Current syphilis
3. Primary language is English or English is a second language but patient self-describes as fluent in English
4. Able to provide informed consent
5. If treated with benzathine penicillin G (BPG), it must have occurred less than 14 days before the entry visit (before the first visit if there is more than one entry visit)

Exclusion Criteria:

1. Provider plans neurosyphilis (NS) treatment regardless of whether the patient has an lumbar puncture (LP)
2. Receipt of antibiotic treatment that would be effective for NS (for example, IV or intramuscular (IM) beta-lactam antibiotics [other than BPG]) within one month before study entry; single dose of IM ceftriaxone in the last month is not exclusionary
3. Allergy to penicillin or lidocaine
4. Contraindication to LP, including untreatable coagulation disorder, use of anticoagulants that cannot be temporarily discontinued, thrombocytopenia, focal neurological examination
5. Other known cause of central nervous system (CNS) infection in the last year, including that due to bacterial, fungal, protozoal or viral agents, such as tuberculosis, Cryptococcus, toxoplasmosis or herpes zoster that could confound interpretation of CSF results
6. Unlikely to be able to comply with study requirements or complete the study, for example, planning to leave the area < 6 months after enrollment
7. Subjects will not be allowed to re-enroll in this study with a new episode of syphilis

Individuals who are unwilling to be randomized can choose LP or no LP. Eligibility criteria for these individuals are:

1. 18 years of age or older
2. Current syphilis infection
3. Primary language is English or fluent in English
4. No contraindications to LP
5. Have not received antibiotics within one month that would treat neurosyphilis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2013-08; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Marra, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol section asks how many participants were enrolled. 219 unique participants were enrolled, but 12 had two enrollments. Thus there are 231 enrollment visits.
Groups:
- Randomized, Lumbar Puncture (LP): Randomized to lumbar puncture (LP) arm
- Reenrolled, Randomized, LP: Randomised after a second enrollment, underwent LP
- Randomized, no LP: Randomized and did not undergo LP. Includes one person for whom LP was unsuccessful.
- Not Randomized, LP: Not randomized and underwent LP.
- Not Randomized, no LP: Not randomized and did not undergo LP.
- Reenrolled, Not Randomized, no LP: Not randomized during another episode of syphilis. Did not undergo LP.
- Reenrolled, Not Randomized, LP: Not randomized with a new episode of syphilis, underwent LP
Period: Overall Study
Arm/Group | Randomized, Lumbar Puncture (LP) | Reenrolled, Randomized, LP | Randomized, no LP | Not Randomized, LP | Not Randomized, no LP | Reenrolled, Not Randomized, no LP | Reenrolled, Not Randomized, LP
Started (There were 231 entry visits for 219 unique individuals. There were 12 re enrollments.) | 11 | 3 | 18 | 148 | 42 | 4 | 5
Considered in Analysis (All participants who were randomized were included in the analysis. The first entry visit for those who were not randomized were included in the analysis if: 1) serum RPR was at or above 1:32 or 2) for PLWH, peripheral blood CD4 + T cells were at or below 350/ul. All included had to have undergone the entry CogState battery.) | 11 | 3 | 18 | 48 | 16 | 0 | 0
Completed (Completed = considered in analysis) | 11 | 3 | 18 | 48 | 16 | 0 | 0
Not Completed | 0 | 0 | 0 | 100 | 26 | 4 | 5
Not completed — Did not meet criteria for inclusion in data analysis | 0 | 0 | 0 | 100 | 26 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Lumbar Puncture Group: Underwent lumbar puncture
- No Lumbar Puncture Group: Did not undergo lumbar puncture
- Total: Total of all reporting groups
Arm/Group | Lumbar Puncture Group | No Lumbar Puncture Group | Total
Number analyzed (Participants) | 62 | 34 | 96
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [29 to 45] | 34 [27 to 40] | 35 [28 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 61 | 34 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants] — number in each category of race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
    Black or African American | 6 | 4 | 10
    White | 45 | 26 | 71
    More than one race | 9 | 1 | 10
    Unknown or Not Reported | 0 | 0 | 0
Serum Rapid Plasma Reagin test (RPR) titer [Median (Inter-Quartile Range); unit: titer] — Titers are expressed as 2-fold dilutions:
  1:1 1:2 1:4 1:8 and so on.
  titer | 128 [32 to 256] | 128 [64 to 256] | 128 [64 to 256]
Impaired on CogState Battery [Number; unit: participants] — The CogState is a computerized battery of neuropsychological tests. Assessment of cognitive impairment was based on age adjusted normative data, categorized as none (all test scores > -1 standard deviation [SD] of normative data), mild impairment (two test scores < -1 SD, or one test score < -2 SD), moderate impairment (two test scores < -2 SD) or severe impairment (three test scores < -2 SD).
  participants | 42 | 20 | 62

OUTCOME MEASURES:

1. Primary Outcome: Appropriate Decline in Serum Rapid Plasma Reagin Test (RPR) Titer
Description: Decline in serum RPR titer by four-fold or to nonreactive at 6 months (+/- 4 weeks) in early syphilis or at 12 months (+/- 4 weeks) in late syphilis. This is the definition of treatment success according to the US Centers for Disease Control and Prevention guidelines.
Time Frame: 6-12 months +/- 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Lumbar Puncture (LP), Treatment Based on Cerebrospinal Fluid (CSF ) Results: Underwent lumbar puncture and treatment based on the results of cerebrospinal fluid findings. Specifically, those with abnormal CSF were treated for neurosyphilis and those without CSF abnormalities were treated for uncomplicated syphilis. The number of participants with late syphilis was too small to allow for separate analysis of early and late stages.
- No Lumbar Puncture Group: Did not undergo lumbar puncture. All were treated for uncomplicated syphilis. The number of participants with late syphilis was too small to allow for separate analysis of early and late stages.
Arm/Group | Lumbar Puncture (LP), Treatment Based on Cerebrospinal Fluid (CSF ) Results | No Lumbar Puncture Group
Number analyzed (Participants) | 42 | 31
Participants | 38 | 30
Statistical Analysis 1: Comparison: Lumbar Puncture (LP), Treatment Based on Cerebrospinal Fluid (CSF ) Results vs No Lumbar Puncture Group; Test type: Other; p = 0.29, Two sample test of proportion in Stata

2. Primary Outcome: Time to Improvement in Performance on CogState Battery.
Description: Assessment of cognitive impairment was based on age adjusted normative data from CogState and was categorized as none (all test scores > -1 standard deviation [SD] of normative data), mild impairment (two test scores < -1 SD, or one test score < -2 SD), moderate impairment (two test scores < -2 SD) or severe impairment (three test scores < -2 SD). Participants were categorized as improved if they had any impairment at study entry and improved by at least one category.
Time Frame: 6-12 months +/- 4 weeks
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Lumbar Puncture (LP), Treatment Based on Cerebrospinal Fluid (CSF ) Results: Underwent lumbar puncture and treatment based on the results of cerebrospinal fluid findings. Specifically, those with abnormal CSF were treated for neurosyphilis and those without CSF abnormalities were treated for uncomplicated syphilis.
- No Lumbar Puncture Group: Did not undergo lumbar puncture. All were treated for uncomplicated syphilis.
Arm/Group | Lumbar Puncture (LP), Treatment Based on Cerebrospinal Fluid (CSF ) Results | No Lumbar Puncture Group
Number analyzed (Participants) | 34 | 20
months | 11.3 [7.5 to 15.2] | 12.2 [3.0 to 21.3]
Statistical Analysis 1: Comparison: Lumbar Puncture (LP), Treatment Based on Cerebrospinal Fluid (CSF ) Results vs No Lumbar Puncture Group; Test type: Other; p = 0.69, Log Rank

3. Post Hoc Outcome: Time to Decline in Performance on the CogState Battery
Description: Participants were categorized as declined if they were not severely impaired at entry and declined by at least one category. The impairment categories are: none (all test scores > -1 standard deviation [SD] of normative data), mild impairment (two test scores < -1 SD, or one test score < -2 SD), moderate impairment (two test scores < -2 SD) or severe impairment (three test scores < -2 SD).
Time Frame: 6-12 months +/- 4 weeks
Population: Time to decline in performance on the CogState battery by log rank test.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Underwent Lumbar Puncture (LP), Abnormal Cerebrospinal Fluid (CSF), Treated for Neurosyphilis (NS): Cerebrospinal fluid (CSF) white cells above 5/ul, supporting the diagnosis of neurosyphilis, and treated for neurosyphilis with antibiotics.
- No LP or Normal CSF and Not Treated for Neurosyphilis: Combination of participants who didn't undergo LP and those who did but had CSF white cells less than or equal to 5/ul and nonreactive cerebrospinal fluid Venereal Disease Research Laboratory (CSF-VDRL) test, and weren't treated for neurosyphilis. In other words, those who didn't undergo LP and those who did have an LP but didn't meet diagnostic criteria for neurosyphilis.
Arm/Group | Underwent Lumbar Puncture (LP), Abnormal Cerebrospinal Fluid (CSF), Treated for Neurosyphilis (NS) | No LP or Normal CSF and Not Treated for Neurosyphilis
Number analyzed (Participants) | 20 | 55
months | NA [NA to NA] — Less than 50% of individuals worsened, so no median time can be reported. | 12.3 [4.1 to 20.5]
Statistical Analysis 1: Comparison: Underwent Lumbar Puncture (LP), Abnormal Cerebrospinal Fluid (CSF), Treated for Neurosyphilis (NS) vs No LP or Normal CSF and Not Treated for Neurosyphilis; Test type: Other; p = 0.04, Log Rank

ADVERSE EVENTS:
Time Frame: One year
Description: No difference
Groups:
- Underwent Lumbar Puncture: Participants who underwent lumbar puncture.
- Did Not Undergo Lumbar Puncture: Participants who did not undergo lumbar puncture.
Arm/Group | Underwent Lumbar Puncture | Did Not Undergo Lumbar Puncture
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/34
Other Adverse Events (participants affected / at risk) | 0/62 | 0/34

LIMITATIONS AND CAVEATS:
Inclusion of a non-randomized group introduces risk of bias; however, the groups were comparable with regard to neurosyphilis risk factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02031146/Prot_SAP_000.pdf